CLINICAL TRIAL: NCT01254305
Title: A Double-blind, Randomized, Placebo- and Active-Controlled Study of F2695 SR in Adult Patients With Fatigue Associated With Major Depressive Disorder
Brief Title: Safety and Efficacy of Levomilnacipran ER (F2695 SR) in Adults With Fatigue Associated With Major Depressive Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LVM-MD-06
Record Dates: First submitted 2010-12-03; First posted 2010-12-06 (Estimated); Results first posted 2014-08-06 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-08

CONDITIONS: Major Depressive Disorder
Keywords: Depression; Fatigue; Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Fatigue | interventions — Levomilnacipran; Paroxetine; Sertraline; Citalopram; Fluoxetine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): 40 -120 mg/day Levomilnacipran ER capsules, oral administration
  Interventions: Drug: Levomilnacipran ER
- 2 (Active Comparator): Randomized to treatment with 1 of 4 Selective Serotonin Reuptake Inhibitors (SSRIs) - Paroxetine, Sertraline, Citalopram or Fluoxetine Oral administration, once daily dosing
  Interventions: Drug: Paroxetine, Sertraline, Citalopram or Fluoxetine.
- 3 (Placebo Comparator): Matching placebo capsules, oral administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levomilnacipran ER — Drug: Levomilnacipran ER (40 -120 mg/day) Study drug is to be given orally, in capsule form, once daily for 8 weeks
  Arms: 1
Drug: Paroxetine, Sertraline, Citalopram or Fluoxetine. — Paroxetine (20, 40, or 60 mg/day) to be given orally, in capsule form, once daily for 8 weeks, or Sertraline (50, 100, or 150 mg/day) to be given orally, in capsule form, once daily for 8 weeks, or Citalopram (20, 40, or 60 mg/day) to be given orally, in capsule form, once daily for 8 weeks or Fluoxetine (20, 40, or 60 mg/day) to be given orally, in capsule form, once daily for 8 weeks
  Arms: 2
Drug: Placebo — Matching placebo capsules, oral administration, once daily dosing
  Arms: 3

SUMMARY:
The purpose of the study is to evaluate the efficacy, safety and tolerability of Levomilnacipran ER for the treatment of fatigue associated with major depressive disorder (MDD).

ELIGIBILITY:
Inclusion Criteria:

* Men and women, 18-65 years old
* Currently meet Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition-Text Revision (DSM-IV-TR) criteria for Major Depressive Disorder
* The patient's current depressive episode must be at least 4 weeks in duration

Exclusion Criteria:

* Women who are pregnant, women who will be breastfeeding during the study, and women of child-bearing potential who are not practicing a reliable method of birth control
* Patients with a history of meeting DSM-IV-TR criteria for:

  1. any manic or hypomanic episode;
  2. schizophrenia or any other psychotic disorder;
  3. obsessive-compulsive disorder.
* Patients who are considered a suicide risk

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2011-04; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carl Gommoll, MS, Study Director — Forest Laboratories
Locations (20):
- United States (20):
  - Forest Investigative Site 010, Birmingham, Alabama
  - Forest Investigative Site 002, Little Rock, Arkansas
  - Forest Investigative Site 001, Cerritos, California
  - Forest Investigative Site 014, Fort Myers, Florida
  - Forest Investigative Site 006, Jacksonville, Florida
  - Forest Investigative Site 017, Orange City, Florida
  - Forest Investigative Site 005, Orlando, Florida
  - Forest Investigative Site 012, Tampa, Florida
  - Forest Investigative Site 009, Atlanta, Georgia
  - Forest Investigative Site 016, Joliet, Illinois
  - Forest Investigative Site 004, New Orleans, Louisiana
  - Forest Investigative Site 022, Boston, Massachusetts
  - Forest Investigative Site 015, Cedarhurst, New York
  - Forest Investigative Site 011, The Bronx, New York
  - Forest Investigative Site 003, Cincinnati, Ohio
  - Forest Investigative Site 013, Dayton, Ohio
  - Forest Investigative Site 020, Lincoln, Rhode Island
  - Forest Investigative Site 018, Memphis, Tennessee
  - Forest Investigative Site 008, Dallas, Texas
  - Forest Investigative Site 007, Middleton, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited over a 12-month period from April of 2011 to April of 2012 at 20 studies sites in the United States.
Pre-assignment Details: Patients went through a 1-week single-blind placebo run-in period, followed by an 8-week double-blind treatment period.
Groups:
- Levomilnacipran ER: 40 -120 mg Levomilnacipran ER capsules, oral administration once daily for 8 weeks.
- SSRI: Randomized to treatment with 1 of 4 Selective Serotonin Reuptake Inhibitors (SSRIs) - Paroxetine, Sertraline, Citalopram or Fluoxetine.
  Paroxetine (20, 40, or 60 mg/day) to be given orally, in capsule form, once daily for 8 weeks, or Sertraline (50, 100, or 150 mg/day) to be given orally, in capsule form, once daily for 8 weeks, or Citalopram (20, 40, or 60 mg/day) to be given orally, in capsule form, once daily for 8 weeks or Fluoxetine (20, 40, or 60 mg/day) to be given orally, in capsule form, once daily for 8 weeks.
Period: Overall Study
Arm/Group | Placebo | Levomilnacipran ER | SSRI
Started | 93 | 90 | 79
Safety Population | 89 | 85 | 77
Completed | 71 | 72 | 62
Not Completed | 22 | 18 | 17
Not completed — Adverse Event | 6 | 3 | 2
Not completed — Lack of Efficacy | 1 | 0 | 1
Not completed — Protocol Violation | 1 | 7 | 3
Not completed — Withdrawal by Subject | 4 | 2 | 4
Not completed — Lost to Follow-up | 10 | 6 | 5
Not completed — Other Reasons | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: A total of 262 patients were randomized to receive double-blind treatment. The Baseline Participant population is based on the 251 randomized patients received at least 1 dose of double-blind treatment (Safety Population).
Groups:
- Placebo: Matching placebo capsules, oral administration
  Placebo : Matching placebo capsules, oral administration, once daily dosing
- Levomilnacipran ER: 40 - 120 mg Levomilnacipran ER capsules, oral administration, once daily for 8 weeks
- Total: Total of all reporting groups
Arm/Group | Placebo | Levomilnacipran ER | SSRI | Total
Number analyzed (Participants) | 89 | 85 | 77 | 251
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.4 (12.0) | 42.9 (12.6) | 42.8 (11.3) | 42.3 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 49 | 49 | 156
  Male | 31 | 36 | 28 | 95
Race/Ethnicity, Customized [Number; unit: participants]
  White | 62 | 57 | 47 | 166
  Black or African American | 26 | 25 | 25 | 76
  Asian | 1 | 3 | 2 | 6
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Other | 0 | 0 | 2 | 2
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 8 | 4 | 10 | 22
  Not Hispanic or Latino | 81 | 81 | 67 | 229
Region of Enrollment [Number; unit: participants]
  United States | 89 | 85 | 77 | 251
Weight [Mean (Standard Deviation); unit: kg] | 79.95 (15.27) | 82.23 (18.14) | 83.31 (17.61) | 81.75 (17.00)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kilograms Per Meter Squared] | 28.16 (4.85) | 28.61 (5.22) | 28.80 (5.10) | 28.51 (5.04)

OUTCOME MEASURES:

1. Primary Outcome: Change in Clinical Global Impression of Severity (CGI-S) for Fatigue Score
Description: The CGI-S is a clinician-rated scale that rates the severity of the patient's current state of fatigue based on the Investigator's clinical opinion with regard to the patient population with Major Depressive Disorder (MDD). Patient were rated on a scale from 1 to 7, with 1 indicating a normal state and 7 indicating that the patient was among the most extremely fatigued
Time Frame: From Baseline to Week 8
Population: The Randomized Population consisted of 262 patients, with 251 patients who took at least 1 dose of double-blind treatment to comprise the Safety population.
  The Intent-to-Treat (ITT) Population consisted of 248 patients in the Safety Population who had a baseline and at least 1 postbaseline assessment of either the CGI-S or PGI-I fatigue score.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo: Dose matched placebo, oral administration in capsule form, once daily for 8 weeks
- Levomilnacipran ER: 40 - 120 mg Levomilnacipran ER capsules, oral administration in capsule form, once daily for 8 weeks
Arm/Group | Placebo | Levomilnacipran ER | SSRI
Number analyzed (Participants) | 88 | 85 | 75
units on a scale | -1.5 (1.3) | -1.8 (1.4) | -1.9 (1.4)

2. Secondary Outcome: Change in Cognitive and Physical Functioning Questionnaire (CPFQ), Last Observation Carried Forward
Description: The Cognitive and Physical Functioning Questionnaire is a patient-rated, 7-item scale used to measure cognitive and executive dysfunction in mood and anxiety disorders. The CPFQ is sensitive to change with treatment and displays convergent validity by significant correlations with other measures of sleepiness, fatigue, apathy, and neuropsychological functioning. Patients are rated on a scale from 1 to 6 for seven common complaints of depressed patients reporting fatigue or cognitive/executive problems-with 1 indicating greater than normal functioning, 2 indicating normal functioning, and 3 to 6 indicating degrees of impaired functioning. The CPFQ ranges from the best possible score of 7 (greater than normal functioning) to the worst possible score of 42 (totally absent).
Time Frame: From Baseline to Week 8
Population: The Randomized Population consisted of 262 patients, with 251 patients who took at least 1 dose of double-blind treatment to comprise the Safety population.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo: Dose matched placebo capsules, oral administration for 8 weeks.
- Levomilnacipran ER: 40 - 120 mg Levomilnacipran ER capsules, oral administration once per day for 8 weeks
Arm/Group | Placebo | Levomilnacipran ER | SSRI
Number analyzed (Participants) | 88 | 85 | 75
units on a scale | -5.9 (7.9) | -7.0 (7.3) | -6.4 (7.0)

3. Primary Outcome: Change in Patient Global Impressions of Severity (PGI-S) for Fatigue Score
Description: The PGI-S is a clinician-rated scale that rates was used to rate the severity of the patient's current state of overall fatigue. Patients were rated on a scale from 1 to 7, with 1 indicating no symptoms of fatigue and 7 indicating extreme fatigue.
Time Frame: From Baseline to Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Levomilnacipran ER | SSRI
Number analyzed (Participants) | 88 | 85 | 75
units on a scale | -1.4 (1.5) | -1.7 (1.5) | -1.7 (1.5)

ADVERSE EVENTS:
Time Frame: Adverse event data occurred over a 16-month period from April of 2011 to September of 2012 at 20 studies sites in the United States.
Description: The Serious Adverse Event data presented here is for the safety population. The Other Adverse Event data presented here is for the safety population during the 8 week double-blind treatment period.
Groups:
- Levomilnacipran ER: 40 -120 mg Levomilnacipran ER capsules, oral administration, once daily for 8 weeks
Arm/Group | Placebo | Levomilnacipran ER | SSRI
Serious Adverse Events (participants affected / at risk) | 0/89 | 1/85 | 0/77
Other Adverse Events (participants affected / at risk) | 39/89 | 41/85 | 37/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=89) | Levomilnacipran ER (N=85) | SSRI (N=77)
Pneumonia (Infections and infestations) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=89) | Levomilnacipran ER (N=85) | SSRI (N=77)
Nausea (General disorders) | 4 | 14 | 6
Headache (Nervous system disorders) | 14 | 12 | 6
Dry mouth (Gastrointestinal disorders) | 6 | 8 | 9
Dizziness (Nervous system disorders) | 2 | 6 | 1
Heart rate increased (Investigations) | 3 | 6 | 0
Diarrhoea (Gastrointestinal disorders) | 8 | 4 | 9
Somnolence (Nervous system disorders) | 4 | 3 | 6
Insomnia (Psychiatric disorders) | 1 | 2 | 5
Anxiety (Psychiatric disorders) | 1 | 1 | 5
Initial insomnia (Psychiatric disorders) | 1 | 1 | 5
Upper respiratory tract infection (Infections and infestations) | 7 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data generated in this study will be the property of Forest Research Institute, Inc. An integrated clinical and statistical report will be prepared at the completion of the study.

Publication of the results by the Investigator will be subject to mutual agreement between the Investigator and Forest Research Institute, Inc.